CLINICAL TRIAL: NCT01184755
Title: RCT of Device-guided Breathing Effects on Ambulatory BP
Brief Title: RCT of Effects of Device-guided Breathing on Ambulatory BP
Acronym: RESPeRate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lynn P. Clemow, Ph.D., ABPP, Clinical Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 526; R01HL083056-01 (NIH)
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Results first posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: Hypertension
Keywords: Device-guided breathing; hypertension; behavioral intervention; stress reduction; Heart Rate Variability (HRV) biofeedback
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resperate device used for 8 weeks (Experimental): Participants to use Resperate device to guide breathing for 8 weeks. After the primary 8-week trial, this group is divided into two subgroups to examine 16-week data: one subgroup that stops using the device after 8 weeks, and one asked to continue to use the device for the full 16 weeks.
  Interventions: Device: RESPeRate
- Relaxation control device (Active Comparator): Participants use modified device to pace breathing in the 13/minute range for daily practice for 8 weeks and no device thereafter
  Interventions: Behavioral: Relaxation
- Usual Care (No Intervention): Participants continue their usual medication and other management for their hypertension. All participants (including UC) are given a home BP monitor and asked to take their BP in morning and evening 3 days/week.

INTERVENTIONS:
Behavioral: Relaxation — Participants are instructed to use the modified device (which paces the breath at a constant 13 breaths/minute) daily for 15 minutes (timing set automatically by device).
  Arms: Relaxation control device
Device: RESPeRate
  Arms: Resperate device used for 8 weeks

SUMMARY:
Our aim is to conduct a randomized controlled trial (RCT) to test the efficacy of a guided breathing intervention on ambulatory blood pressure (ABP), both systolic and diastolic BP. There are 3 groups: 1) Intervention group instructed to use the RESPeRate device that guides the breath into the 6 breaths/minute range daily for 8 weeks. 2) Relaxation control condition (using a modified device to guide breathing at 13 breaths/minute rate); and 3) Usual Care (UC). After the initial 8 week trial, the main outcome, the intervention group will be randomly assigned to stop using the RESPeRate device or to continue using it for 8 more weeks.

DETAILED DESCRIPTION:
Device-guided breathing is a behavioral intervention that guides the breathing into the 6 per minute range, inducing respiratory sinus arrythmia (RSA), which is the natural cycle of arrythmia that occurs through the influence of breathing on the flow of sympathetic and vagus impulses to the sinoatrial node of the heart. It has been shown in several small trials to have substantial effects on BP reduction, has no known side-effects, and may represent a cost-effective adjunctive treatment for hypertension. an important consideration is that, often, behavioral interventions are given for a brief amount of time, but are expected to have long-term effects. This does not hold true for medication; one would not give anti-hypertensive medication for eight weeks and expect an effect on BP several months later. The development of behavioral interventions needs to take into account methods to sustain long-term effects.

Our aim is to conduct a randomized controlled trial (RCT) to test the efficacy of a guided breathing intervention on ambulatory BP (ABP) in hypertensives drawn from primary care and specialty hypertension practices, using a sample size powered to detect effects at 8 weeks and 4-month follow-up. The design calls for two control groups: Usual Care (UC) and a relaxation control condition (using a device that gives the same type of feedback sounds as the guided breathing feedback device, but modified to pace the breathing at approximately 13 breaths per minute, a normal resting rate.) The intervention condition has participants use the RESPeRate device that guides the breath into the 6 breaths/minute range. The initial intervention lasts eight weeks, following which participants are further randomized to either: 1) ending the intervention; of 2) continuing the intervention for the next 8 weeks. The main outcomes are the change at 8 weeks in systolic and diastolic BP (measured by Ambulatory BP monitoring) during the waking hours. Outcomes are measured at baseline, 8 weeks, and 16 weeks. The primary outcomes are BP results at 8 weeks, with a 3-group comparison of the intervention group, the relaxation control group and usual care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hypertension
* Treated with at least one antihypertensive drug
* BP still not controlled (>135/85 on Ambulatory BP waking average)

Exclusion Criteria:

* Diabetes
* Atrial Fibrillation
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2008-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn P Clemow, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Resperate Device Used for 8 Weeks: Participants to use Resperate device to guide breathing for 8 weeks, then not used for next 8 weeks
  Device-guided breathing: Participants instructed to practice daily for 15 minutes (guided and timed by the device used at home)
  RESPeRate
- Relaxation Placebo Device: Participants use modified device to pace breathing in the 13/minute range for daily practice for 8 weeks and no device thereafter
  Relaxation: Participants are instructed to use the device (which paces the breath at a constant 13 breaths/minute) daily for 15 minutes (timing set automatically by device).
  Sham RESPeRate
Period: Overall Study
Arm/Group | Resperate Device Used for 8 Weeks | Relaxation Placebo Device | Usual Care
Started | 126 | 65 | 62
Completed | 101 | 54 | 56
Not Completed | 25 | 11 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resperate Device Used for 8 Weeks | Relaxation Placebo Device | Usual Care | Total
Number analyzed (Participants) | 126 | 65 | 62 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 101 | 51 | 51 | 203
  >=65 years | 25 | 14 | 11 | 50
Age, Continuous [Mean (Full Range); unit: years] | 56.65 [23 to 80] | 57.58 [34 to 79] | 56.34 [27 to 76] | 56.74 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 33 | 34 | 138
  Male | 55 | 32 | 28 | 115
Region of Enrollment [Number; unit: participants]
  United States | 126 | 65 | 62 | 253

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic and Diastolic BP Measured by Ambulatory BP Monitoring (Waking Averages)
Description: The primary outcome for this study is the change in systolic and diastolic BP measured by Ambulatory BP monitoring at 8-weeks. The measure is the waking mean BP.
Time Frame: 8 weeks
Population: These were patients who completed both the baseline and 8-week Ambulatory BP measures.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Resperate Device Used for 8 Weeks | Relaxation Placebo Device | Usual Care
Number analyzed (Participants) | 101 | 54 | 56
mm Hg
  Change in Systolic BP | 5.8 (10.7) | 6.6 (12.3) | 1.2 (9.9)
  Change in Diastolic BP | 4.0 (7.0) | 4.7 (7.4) | 0.5 (7.1)
Statistical Analysis 1: Comparison: Resperate Device Used for 8 Weeks vs Relaxation Placebo Device vs Usual Care; This is the change in Systolic BP at 8 weeks; Test type: Superiority or Other; p = .01, Mixed effects regression analysis — This is an intention-to-treat analysis; Mean Difference (Final Values) = -.561256, 95% CI 2-sided [-.987999 to -.134513], Standard Error of Mean .216403
Statistical Analysis 2: Comparison: Resperate Device Used for 8 Weeks vs Relaxation Placebo Device vs Usual Care; This is the analysis of change in diastolic BP from Ambulatory BP monitoring; Test type: Superiority or Other; p = .006, mixed effects regression analysis; Mean Difference (Final Values) = -.391195, 95% CI 2-sided [-.667312 to -.115079], Standard Error of Mean .140034

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: This was the duration of their participation in the study.
Arm/Group | Resperate Device Used for 8 Weeks | Relaxation Placebo Device | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/126 | 0/65 | 0/62
Other Adverse Events (participants affected / at risk) | 0/126 | 0/65 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No